CLINICAL TRIAL: NCT06543979
Title: The Diagnostic Value of Anorectal Manometry in Pediatric Chronic Refractory Constipation With or Without Fecal Incontinence
Brief Title: Anorectal Manometery in Pediatric Chronic Refractory Constipation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, asmaa abdelnaby, assistant lecturer of pediatrics, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: manometery in constipation
Record Dates: First submitted 2024-05-09; First posted 2024-08-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — Lubiprostone; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- single arm as all participant will receive the treatment (Other): all participant will receive lubiprostone
  Interventions: Drug: lubiprostone , single arm; Procedure: biofeed back sessions; Procedure: botox injection

INTERVENTIONS:
Drug: lubiprostone , single arm — laxative
  Other Names: lubicont
Procedure: biofeed back sessions — Biofeedback for participants with dyssynergic defecation and participants with reduced rectal sensations
Procedure: botox injection — Botulinum toxin injection for participants suffering from elevated anal canal pressure

SUMMARY:
Anorectal manometry and high-resolution anorectal manometry (HRAM) are becoming the investigation of choice for understanding the pathophysiology of chronic constipation with or without fecal incontenance in children in many institutions. In high resolution anorectal manometery we are able to gain information whether the symptoms are related to sphincter dysfunction, impaired sensation, or pelvic floor dyssynergia

DETAILED DESCRIPTION:
Primary objective: To assess different patterns of anorectal manometry in children with chronic refractory constipation with or without fecal incontinence.

Secondary objective: To determine the effectiveness of different modalities of treatment of chronic refractory constipation based on the anorectal findings. To assess the safety ,tolerability and effectiveness of lubiprostone in pediatric age group with chronic refractory constipation. To assess the effect of elimination of cow milk products in patient with chronic refractory constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents aged from 4 to 16 years.
2. Participants fulfilling Rome IV criteria for the diagnosis of functional constipation.

   At least 2 of the following present at least once per week for at least 1 month:
   * 2 or fewer defecations in the toilet per week
   * At least 1 episode of fecal incontinence per week
   * History of retentive posturing or excessive volitional stool retention
   * History of painful or hard bowel movements
   * Presence of a large fecal mass in the rectum
   * History of large-diameter stools that may obstruct the toilet The symptoms cannot be fully explained by another medical condition (Hyams et al., 2016).
3. Participants who have chronic refractory constipation. Chronic refractory constipation (CRC) is defined as children who are unable to pass stools in spite of being on maximum laxative therapy and require daily rectal stimulation in the form of enemas or suppositories to pass stools 4-Is willing and able to keep a diary on his/her own and willing and able to complete a questionnaire.

5-The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.

Exclusion Criteria:

* participants who have anorectal malformation
* participants who have neurological disease affecting lower limbs
* Has a history of hypersensitivity or allergies to lubiprostone

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-07 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the manometric parameters in children with chronic refractory constipation | 1 year
  To measure the percent of the most common manometric parameters in children with chronic refractory constipation e.g dyssengeric defecation and reduced rectal sensetivity and anal sphincter dysfunction.
evaluate the efficacy of oral administration of lubiprostone 8 and 24 μg once daily for 4 weeks in participants with chronic refractory constipation | 1 month
  Spontaneous Bowel Movement (SBM) Frequency at Week 1,2,3 and 4 A SBM was defined as any bowel movement (BM) that does not occur within 24 hours after rescue medication use (laxative, suppository, or enema). Participants will be given a diary to complete at home where they will record all details of each SBM including the consistency of the stool and the difficulty they have in passing it.

SECONDARY OUTCOMES:
To determine the effect of biofeed back sessions in children with dyssengeric defecation and in children with rectal hyposensetivity | 3 months
  Participants with chronic refractory constipation and manometry parameters showed dyssengeric defecation or hyposensitivity will receive biofeedback sessions and the investigators measure the difference in bowel management scoring tool before and after the biofeedback sessions the higher the score the worest the condition
To determine the effect of cow milk protein free diet on chronic refractory constipation in children | 1 month
  Participants will receive cow milk free diet for 4 weeks and investigators measure the difference in bowel management scoring tool before and after cow milk free diet the higher the score the worest the condition
To determine the effect of botulinum toxin injection in children with elevated anal canal resting pressure | 3 month
  Participants with chronic refractory and manometric parameters showed high anal canal resting pressure will have botulinum toxin injection and investigators measure the difference in bowel management scoring tool before and after the injection the higher the score the worest the condition

CONTACTS AND LOCATIONS:
Overall Officials: asmaa abdelnaby mohamed soliman, master, Principal Investigator — assistant lecturer
Locations (1):
- Ain shams university, Cairo, Egypt